CLINICAL TRIAL: NCT04882657
Title: Collateral Circulation ("Collaterome") in Acute Ischemic Stroke With Large Vessel Occlusion: A Study of Clinical, Radiological, Plasma and Genetic Factors.
Brief Title: Collateral Circulation in Acute Ischemic Stroke With Large Vessel Occlusion
Acronym: COLISEUM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Complejo Hospitalario Universitario de Albacete (Other); Hospital de Cruces (Other); Hospital Clínico Universitario de Valladolid (Other); Hospitales Universitarios Virgen del Rocío (Other); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Hospital Universitario La Paz (Other); Hospital del Mar (Other); Hospital Arnau de Vilanova (Other); Complexo Hospitalario Universitario de A Coruña (Other); Red de Enfermedades Vasculares Cerebrales INVICTUS PLUS (Rd1600190024) (Unknown)
Responsible Party: Sponsor
Other Study IDs: IIBSP-COL-2019-64
Record Dates: First submitted 2019-12-05; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Stroke, Ischemic; Stroke, Acute; Collateral Circulation, Any Site
Keywords: Collateral Circulation; Ischemic Stroke; Large Vessel Occlusion
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sampling will be obtained by venipuncture in EDTA tubes at admission and processed at each center. Samples will be sent to the promoter site for genetic and plasma markers analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective multicenter study of consecutive patients with acute ischemic stroke and large intracranial vessel occlusion in which a thorough and systematic evaluation of all variables that may be related to the degree of collateral circulation is performed.

DETAILED DESCRIPTION:
Introduction. In patients with an acute ischemic stroke due to a large-vessel intracranial occlusion (LVO), the status of the colateral circulation (CC) is related to clinical outcome and to the success of mechanical thrombectomy. However, CC is highly variable from patient to patient.

Methods. An observational, prospective, multicenter study of 700 consecutive patients with acute ischemic stroke and a LVO. Factors to be evaluated: 1) Modifiable: Vascular risk factors, blood analysis, prior medications, vital constants (with emphasis on continuous blood pressure monitoring), head position, metrics (time to admission, Computed tomography (CT), groin puncture, end of procedure), 2) Non-modifiable: age, sex, completeness of Circle of Willis, etiology, type of mechanical thrombectomy, plasma biomarkers, genetic/epigenetic factors (a discovery phase with GWAs study and a replication phase). CC grade will be assessed by the ASITN/SIR collateral score from CT-angiography (CTA) and the Digital substraction angiography (DSA, when performed). Statistics: bivariate analyses and a logistic regression to predict CC grade (poor versus good) and CC persistence comparing CTA with DSA (4 possibilities: poor-poor, poor-good, good-poor, good-good).

Expected results. Our study may find markers of the CC status, facilitate the design of clinical trials to improve CC grade, may find new therapeutic targets and new treatments to enhance the beneficial effects of mechanical thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke.
* Large vessel occlusion of an intracranial internal artery: M1, M2 or TICA. (terminal intracranial carotid artery), as demonstrated by CTA.
* CTA performed within the first 24 hours after stroke onset. Patients with wake-up stroke are included.
* A previous modified Rankin Scale score of 0 to 3.
* The patient or a legal representative signs a written consent to participate.

Exclusion Criteria:

* More than 24 hours from last been known to be well.
* Occlusion of other arterial segments (vertebrobasilar circulation, A1, P1, M3, M4).
* Age below 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke and a large-vessel intracranial occlusion.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Collateral Circulation grade | Trough the acute phase of stroke, an average of 24 hours

IPD SHARING:
Plan to Share IPD: Undecided